CLINICAL TRIAL: NCT02954458
Title: A Prospective, Open-label, Long-term Safety and Efficacy Study of Teduglutide in Pediatric Patients With Short Bowel Syndrome Who Completed TED-C14-006 or SHP633-301
Brief Title: Long-term Safety and Efficacy Study of Teduglutide in Pediatric Participants With Short Bowel Syndrome (SBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-304; 2016-000849-30 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Syringes; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Standard of care (SOC) treatment +/- teduglutide (TED) (Experimental): Participants will receive 0.05 milligram per kilogram (mg/kg) of teduglutide subcutaneous (SC) injections once daily into 1 of the 4 quadrants of the abdomen or into either the thigh or arm as needed in addition to SOC treatment.
  Interventions: Drug: TED; Other: SOC; Device: Syringe; Device: Needle

INTERVENTIONS:
Drug: TED — 0.05 mg/kg SC injection once daily.
Other: SOC — Standard safety assessments and adjustments in nutritional support.
Device: Syringe — Teduglutide will be administered using syringe.
Device: Needle — Teduglutide will be administered using needle.

SUMMARY:
This study will follow participants who completed the TED-C14-006 study. The purpose of this study is to evaluate the long-term safety and efficacy of teduglutide in pediatric participants with Short Bowel Syndrome (SBS). This study will also offer teduglutide treatment to eligible participants, regardless of treatment received in TED-C14-006 or SHP633-301.

ELIGIBILITY:
Inclusion Criteria:

1. Participant provides written informed consent (participant, parent or legal guardian and, as appropriate, informed assent) to participate in the study before completing any study-related procedures.
2. Participant completed the TED-C14-006 or SHP633-301 studies (including participants in the standard of care treatment arms). Participants are considered to have completed SHP633-301 if they completed study assessments through week 24.
3. Participant understands and is willing and able to fully adhere to study requirements as defined in this protocol.

Exclusion Criteria:

1. There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (22):
- United States (15):
  - Childrens Hospital Los Angeles - RHU, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Georgetown Children's Research Network, Washington D.C., District of Columbia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - The Nebraska Medical Center, Omaha, Nebraska
  - Columbia Unversity Medical Center, New York, New York
  - Children's Hosp. at Montefiore, The Bronx, New York
  - Duke Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Cliniques Universitaires Saint-Luc, Brussels, Woluwe-Saint-Lambert, Belgium
- Canada (2):
  - Walter C. Mackenzie Health Science Centre, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
- Helsingin yliopistollinen keskussairaala, Helsinki, Finland
- Ospedale Pediatrico Bambino Gesu, Roma, Italy
- United Kingdom (2):
  - Great Ormond Children's Hosp, London, Greater London
  - Birmingham Children's Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab470c2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 sites between 09 January 2017 and 05 November 2020. A total of 61 participants (children and infant) were enrolled and classified into treatment groups (NTT/NTT, NTT/TED , TED/NTT, and TED/TED) based on whether they received teduglutide in their core study TED-C14-006 [NCT02682381] or SHP633-301 [NCT03571516] and/or during this extension study. Participants who completed their core study were eligible for this extension study.
Pre-assignment Details: NTT/NTT: Participants who participated in standard of care (SOC) arm in the core study and didn't receive any TED treatment in this extension study; NTT/TED: Participants who participated in SOC arm in the core study but who subsequently received TED in this extension study; TED/NTT: Participants who received TED in the core study but didn't receive any TED treatment in this extension study; TED/TED: Participants who received TED in the core study and in this extension study.
Groups:
- Non-teduglutide/Non-teduglutide Treatment (NTT/NTT): Participants who participated in standard of care arm in the core study TED-C14-006 [NCT02682381] or SHP633-301 [NCT03571516] were enrolled into this extension study but did not receive any teduglutide treatment in this extension study.
- Non-teduglutide/Teduglutide Treatment (NTT/TED): Participants who participated in standard of care arm in the core study TED-C14-006 [NCT02682381] or SHP633-301 [NCT03571516] were enrolled into this extension study and received 0.05 milligram per kilogram (mg/kg) of teduglutide subcutaneous (SC) injections once daily up to 121 weeks.
- Teduglutide /Non-teduglutide Treatment (TED/NTT): Participants who received teduglutide in the core study TEDC14-006 [NCT02682381] or SHP633-301 [NCT03571516] were enrolled into this extension study but did not receive any teduglutide treatment in this extension study.
- Teduglutide/Teduglutide Treatment (TED/TED): Participants who received teduglutide in the core study TED-C14-006 [NCT02682381] or SHP633-301 [NCT03571516] were enrolled into this extension study received 0.05 mg/kg of teduglutide SC injections once daily up to 142 weeks.
Period: Overall Study
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Started | 7 | 3 | 1 | 50
Completed | 6 | 3 | 0 | 38
Not Completed | 1 | 0 | 1 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: The safety population consisted of enrolled participants who provided informed consent and met all the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED) | Total
Number analyzed (Participants) | 7 | 3 | 1 | 50 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.8 (5.43) | 1.5 (0.80) | 6.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 5.7 (3.69) | 5.5 (3.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 16 | 20
  Male | 4 | 2 | 1 | 34 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 0 | 1 | 38 | 42
  Race: Black or African American | 1 | 0 | 0 | 6 | 7
  Race: Asian | 1 | 1 | 0 | 1 | 3
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Other | 1 | 1 | 0 | 1 | 3
  Race: Not allowed based on local regulations | 1 | 1 | 0 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 1 | 0 | 10 | 14
  Ethnicity: Not Hispanic or Latino | 3 | 1 | 1 | 35 | 40
  Ethnicity: Not allowed based on local regulations | 1 | 1 | 0 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that started or worsened on or after the date of first dose of teduglutide for participants in the TED/TED, TED/NTT, and NTT/TED treatment groups, or after the core study baseline visit for participants in the NTT/NTT group.
Time Frame: From start of study drug administration up to follow-up (up to 46 months)
Population: The safety population consisted all enrolled participants who provided informed consent and met all the inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 7 | 3 | 1 | 50
Participants | 6 | 3 | 1 | 50

2. Primary Outcome: Change From Baseline in Average Total Urine Output at End of Treatment (EOT) of Last Cycle During Teduglutide Treatment
Description: Average total urine output was recorded over a 48-hour period of parental support (PS) stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The Average daily urine output milliliter per kilogram per day (mL/kg/day) was calculated as: Total urine output over 48 hours / 2) / body weight (kilogram [kg]) where total urine output was calculated as the sum of the urine output in milliliter (mL) and the urine-only diaper weights in gram (g) (1g = 1mL) for the participant collected on the output diary form of electronic case report from (eCRF).
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: The safety population consisted all enrolled participants who provided informed consent and met all the inclusion criteria. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure. Data was collected and analyzed for NTT/TED, and TED/TED arms in Teduglutide treatment.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 32
mL/kg/day | 0.26 (1.692) | 2.51 (22.607)

3. Primary Outcome: Change From Baseline in Average Total Urine Output at Last Visit During Non-Teduglutide Treatment (NT)
Description: Average total urine output was recorded over a 48 hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. Average daily urine output mL/kg/day was calculated as: (Total urine output over 48 hours/2) / body weight (kg) where total urine output was calculated as the sum of the urine output in mL and the urine-only diaper weights in gram (1g = 1mL) for the participant collected on the output diary form of electronic case report from (eCRF).
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: The safety population consisted all enrolled participants who provided informed consent and met all the inclusion criteria. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure. Data was collected and analyzed for all the four arms: NTT/NTT, NTT/TED, TED/NTT and TED/TED. Participants who received teduglutide treatment could enter a NT period when the teduglutide treatment criteria were not met.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 4 | 0 | 1 | 11
mL/kg/day | -0.89 (7.431) |  | 15.01 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -6.87 (26.299)

4. Primary Outcome: Change From Baseline in Average Number of Stools Per Day at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized by the average number of stools per day. The average number of stools per day was calculated as (sum of the daily data in a 48-hour period/2).
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Stools per day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 0 | 32
Stools per day |  | -0.47 (2.272)

5. Primary Outcome: Change From Baseline in Average Number of Stools Per Day at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 4
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Stools per day
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 4 | 0 | 0 | 14
Stools per day | -0.50 (0.913) |  |  | 0.38 (1.780)

6. Primary Outcome: Change From Baseline in Average Total Daily Stool/Mixed Stool Diaper Weight at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized by the average total daily stool/mixed stool diaper weight (gram per kilogram per day [g/kg/day]). The body weight was used to calculate the daily stool/mixed stool diaper weight (g/kg/day).
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 1 | 7
g/kg/day | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -11.35 (25.667)

7. Primary Outcome: Change From Baseline in Average Total Daily Stool/Mixed Stool Diaper Weight at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 6
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 1 | 0 | 0 | 4
g/kg/day | 0.31 (NA) — Standard deviation could not be calculated because single participant was analyzed. |  |  | -4.98 (20.892)

8. Primary Outcome: Change From Baseline in Average Total Ostomy Output at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized the average ostomy output per day (mL/kg/day).
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 5
mL/kg/day | -12.52 (11.675) | 12.16 (35.079)

9. Primary Outcome: Change From Baseline in Average Total Ostomy Output at Last Visit During Non-Teduglutide Treatment (NT)
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized the average ostomy output per day.
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 0 | 0 | 0 | 2
mL/kg/day |  |  |  | 23.89 (37.835)

10. Primary Outcome: Change From Baseline in Average Bristol Stool Form Score at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The Average daily fecal output was summarized the average typical stool form score using Bristol Stool Form Scale. The average typical stool form score was calculated as (sum of the daily data in a 48-hour period / 2). Typical Stool Form based on Bristol Stool Form Scale: 1 - Separate hard lumps, hard to pass, 2 - Sausage-shaped, but lumpy, 3 - Like a sausage but with cracks on the surface, 4- Like a sausage or snake, smooth and soft, 5- Soft blobs with clear-cut edges, 6- Fluffy pieces with ragged edges, a mushy stool, 7- Watery, no solid pieces. Entirely liquid.
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scale on a Score
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 0 | 32
Scale on a Score |  | -0.54 (0.977)

11. Primary Outcome: Change From Baseline in Average Bristol Stool Form Score at Last Visit During Non-Teduglutide Treatment (NT)
Description: Fecal output was recorded over a 48 hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized separately the average typical stool form score using Bristol Stool Form Scale. The average typical stool form score was calculated as (sum of the daily data in a 48-hour period / 2). Typical Stool Form based on Bristol Stool Form Scale: 1- Separate hard lumps, hard to pass, 2- Sausage-shaped, but lumpy, 3- Like a sausage but with cracks on the surface, 4 - Like a sausage or snake, smooth and soft, 5- Soft blobs with clear-cut edges, 6- Fluffy pieces with ragged edges, a mushy stool, 7- Watery, no solid pieces. Entirely liquid.
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scale on a Score
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 4 | 0 | 1 | 14
Scale on a Score | -0.25 (0.500) |  | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -0.08 (0.583)

12. Primary Outcome: Number of Participants With Positive Specific Antibodies at End of Study (EOS)
Description: Number of participants with positive specific antibodies to teduglutide were used to summarize the presence of antibodies.
Time Frame: At EOS (up to 46 months)
Population: The safety population consisted all enrolled participants who provided informed consent and met all the inclusion criteria. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure. Data was collected and analyzed for the 3 arms: NTT/TED, TED/NTT and TED/TED only.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 1 | 40
Participants | 2 | 0 | 10

13. Primary Outcome: Change From Baseline in Body Weight Z-score at EOT of Last Cycle During Teduglutide Treatment
Description: Body weight was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 43
Z-score | 0.087 (0.422) | -0.164 (0.951)

14. Primary Outcome: Change From Baseline in Body Weight Z-score at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 13
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 1 | 1 | 19
Z-score | -0.489 (0.542) | -0.132 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 0.013 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -0.363 (0.657)

15. Primary Outcome: Change From Baseline in Height Z-score at EOT of Last Cycle During Teduglutide Treatment
Description: Height was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 27
Z-score | 0.118 (0.968) | -0.277 (0.797)

16. Primary Outcome: Change From Baseline in Height Z-score at Last Visit During Non-Teduglutide Treatment
Description: as for outcome 15
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 1 | 1 | 18
Z-score | -0.518 (0.451) | -0.770 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 0.220 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -0.132 (0.466)

17. Primary Outcome: Change From Baseline in Head Circumference Z-score at EOT of Last Cycle During Teduglutide Treatment
Description: Head circumference was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 0 | 2
Z-score |  | -0.727 (0.440)

18. Primary Outcome: Change From Baseline in Head Circumference Z-score at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 17
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 0 | 0 | 0 | 1
Z-score |  |  |  | -0.309 (NA) — Standard deviation could not be calculated because single participant was analyzed.

19. Primary Outcome: Change From Baseline in Body Mass Index (BMI) Z-score at EOT of Last Cycle During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight data. Z-score was calculated as (observed value - median value of the reference population) / standard deviation value of reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts are used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline, EOT of last cycle (up to Month 36) (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 43
Z-score | 0.215 (0.142) | 0.035 (0.904)

20. Primary Outcome: Change From Baseline in Body Mass Index (BMI) Z-score at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 19
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 1 | 1 | 19
Z-score | -0.545 (1.335) | 0.791 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -0.564 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -0.148 (0.555)

21. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%), 50%, and 75% Reduction From Baseline in Diary Parenteral Support (PS) Volume at End of Treatment (EOT) of Each Cycle During Teduglutide Treatment
Description: Number of participants who achieved at least 20%, 50%, and 75% reduction from baseline in diary PS volume at EOT of last cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: The safety population consisted all enrolled participants who provided informed consent and met all the inclusion criteria. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. Data was collected and analyzed for NTT/TED, and TED/TED arms in Teduglutide treatment. Number of participants in each categories are mutually exhaustive at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
Participants
  Change at EOT of Cycle 1: >= 20% Reduction | 1 | 29
  Change at EOT of Cycle 1: >= 50% Reduction | 0 | 13
  Change at EOT of Cycle 1: >= 75% Reduction | 0 | 7
  Change at EOT of Cycle 2: >= 20% Reduction: number analyzed (Participants) | 2 | 43
  Change at EOT of Cycle 2: >= 20% Reduction | 1 | 29
  Change at EOT of Cycle 2: >= 50% Reduction: number analyzed (Participants) | 2 | 43
  Change at EOT of Cycle 2: >= 50% Reduction | 0 | 17
  Change at EOT of Cycle 2: >= 75% Reduction: number analyzed (Participants) | 2 | 43
  Change at EOT of Cycle 2: >= 75% Reduction | 0 | 9
  Change at EOT of Cycle 3: >= 20% Reduction: number analyzed (Participants) | 2 | 33
  Change at EOT of Cycle 3: >= 20% Reduction | 2 | 22
  Change at EOT of Cycle 3: >= 50% Reduction: number analyzed (Participants) | 2 | 33
  Change at EOT of Cycle 3: >= 50% Reduction | 0 | 14
  Change at EOT of Cycle 3: >= 75% Reduction: number analyzed (Participants) | 2 | 33
  Change at EOT of Cycle 3: >= 75% Reduction | 0 | 6
  Change at EOT of Cycle 4: >= 20% Reduction: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4: >= 20% Reduction | 1 | 20
  Change at EOT of Cycle 4: >= 50% Reduction: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4: >= 50% Reduction | 1 | 13
  Change at EOT of Cycle 4: >= 75% Reduction: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4: >= 75% Reduction | 0 | 7
  Change at EOT of Cycle 5: >= 20% Reduction: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5: >= 20% Reduction | 1 | 15
  Change at EOT of Cycle 5: >= 50% Reduction: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5: >= 50% Reduction | 1 | 13
  Change at EOT of Cycle 5: >= 75% Reduction: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5: >= 75% Reduction | 0 | 6
  Change at EOT of Cycle 6: >= 20% Reduction: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6: >= 20% Reduction | 0 | 2
  Change at EOT of Cycle 6: >= 50% Reduction: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6: >= 50% Reduction | 0 | 2
  Change at EOT of Cycle 6: >= 75% Reduction: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6: >= 75% Reduction | 0 | 1
  Change at EOT of Last Cycle: >= 20% Reduction | 3 | 29
  Change at EOT of Last Cycle: >= 50% Reduction | 1 | 21
  Change at EOT of Last Cycle: >= 75% Reduction | 0 | 11

22. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%), 50%, and 75% Reduction From Baseline in Prescribed PS Volume at End of Treatment (EOT) of Each Cycle During Teduglutide Treatment
Description: Number of participants who achieved at least 20%, 50%, and 75% reduction from baseline in prescribed PS volume at EOT of east cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: The safety population consisted all enrolled participants who provided informed consent and met all the inclusion criteria. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. Data was collected and analyzed for NTT/TED, and TED/TED arms in Teduglutide treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
Participants
  EOT of Cycle 1: >= 20% Reduction in PS Volume | 2 | 35
  EOT of Cycle 1: >= 50% Reduction in PS Volume | 0 | 18
  EOT of Cycle 1: >= 75% Reduction in PS Volume | 0 | 9
  EOT of Cycle 2: >= 20% Reduction in PS Volume: number analyzed (Participants) | 2 | 43
  EOT of Cycle 2: >= 20% Reduction in PS Volume | 2 | 31
  EOT of Cycle 2: >= 50% Reduction in PS Volume: number analyzed (Participants) | 2 | 43
  EOT of Cycle 2: >= 50% Reduction in PS Volume | 2 | 18
  EOT of Cycle 2: >= 75% Reduction in PS Volume: number analyzed (Participants) | 2 | 43
  EOT of Cycle 2: >= 75% Reduction in PS Volume | 1 | 11
  EOT of Cycle 3: >= 20% Reduction in PS Volume: number analyzed (Participants) | 2 | 33
  EOT of Cycle 3: >= 20% Reduction in PS Volume | 2 | 24
  EOT of Cycle 3: >= 50% Reduction in PS Volume: number analyzed (Participants) | 2 | 33
  EOT of Cycle 3: >= 50% Reduction in PS Volume | 1 | 14
  EOT of Cycle 3: >= 75% Reduction in PS Volume: number analyzed (Participants) | 2 | 33
  EOT of Cycle 3: >= 75% Reduction in PS Volume | 1 | 7
  EOT of Cycle 4: >= 20% Reduction in PS Volume: number analyzed (Participants) | 1 | 27
  EOT of Cycle 4: >= 20% Reduction in PS Volume | 1 | 21
  EOT of Cycle 4: >= 50% Reduction in PS Volume: number analyzed (Participants) | 1 | 27
  EOT of Cycle 4: >= 50% Reduction in PS Volume | 1 | 13
  EOT of Cycle 4: >= 75% Reduction in PS Volume: number analyzed (Participants) | 1 | 27
  EOT of Cycle 4: >= 75% Reduction in PS Volume | 0 | 7
  EOT of Cycle 5: >= 20% Reduction in PS Volume: number analyzed (Participants) | 1 | 20
  EOT of Cycle 5: >= 20% Reduction in PS Volume | 1 | 17
  EOT of Cycle 5: >= 50% Reduction in PS Volume: number analyzed (Participants) | 1 | 20
  EOT of Cycle 5: >= 50% Reduction in PS Volume | 1 | 12
  EOT of Cycle 5: >= 75% Reduction in PS Volume: number analyzed (Participants) | 1 | 20
  EOT of Cycle 5: >= 75% Reduction in PS Volume | 0 | 6
  EOT of Cycle 6: >= 20% Reduction in PS Volume: number analyzed (Participants) | 0 | 3
  EOT of Cycle 6: >= 20% Reduction in PS Volume |  | 2
  EOT of Cycle 6: >= 50% Reduction in PS Volume: number analyzed (Participants) | 0 | 3
  EOT of Cycle 6: >= 50% Reduction in PS Volume |  | 2
  EOT of Cycle 6: >= 75% Reduction in PS Volume: number analyzed (Participants) | 0 | 3
  EOT of Cycle 6: >= 75% Reduction in PS Volume |  | 0
  EOT of Last Cycle: >= 20% Reduction in PS Volume | 3 | 37
  EOT of Last Cycle: >= 50% Reduction in PS Volume | 2 | 23
  EOT of Last Cycle: >= 75% Reduction in PS Volume | 1 | 12

23. Secondary Outcome: Change From Baseline in Diary PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in diary PS volume at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
mL/kg/day
  Change at EOT of Cycle 1 | -14.87 (4.574) | -22.63 (18.125)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Change at EOT of Cycle 2 | -8.98 (10.490) | -25.75 (22.480)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Change at EOT of Cycle 3 | -34.81 (15.314) | -32.01 (28.837)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Change at EOT of Cycle 4 | -57.45 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -32.61 (24.639)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Change at EOT of Cycle 5 | -56.90 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -38.76 (21.148)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -40.51 (24.833)
  Change at EOT of Last Cycle | -33.39 (20.503) | -29.36 (25.514)

24. Secondary Outcome: Percent Change From Baseline in Diary PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in diary PS volume at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
Percent change
  Percent Change at EOT of Cycle 1 | -23.23 (15.103) | -41.88 (34.100)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Percent Change at EOT of Cycle 2 | -13.29 (16.826) | -45.67 (38.377)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Percent Change at EOT of Cycle 3 | -38.66 (2.603) | -46.62 (37.756)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Percent Change at EOT of Cycle 4 | -50.99 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -51.28 (36.364)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Percent Change at EOT of Cycle 5 | -50.50 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -58.86 (33.522)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -52.87 (32.722)
  Percent Change at EOT of Last Cycle | -42.65 (7.061) | -50.27 (38.917)

25. Secondary Outcome: Change From Baseline in Prescribed PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in prescribed PS volume at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
mL/kg/day
  Change at EOT of Cycle 1 | -22.57 (13.957) | -20.87 (20.957)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 43
  Change at EOT of Cycle 2 | -65.88 (12.621) | -24.24 (24.914)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 33
  Change at EOT of Cycle 3 | -58.82 (4.022) | -30.53 (26.449)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4 | -68.72 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -34.53 (23.849)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5 | -68.99 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -37.78 (22.850)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -39.10 (24.154)
  Change at EOT of Last Cycle | -48.23 (25.528) | -26.26 (25.275)

26. Secondary Outcome: Percent Change From Baseline in Prescribed PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: Percent Change from baseline in prescribed PS volume at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
Percent Change
  Percent Change at EOT of Cycle 1 | -28.82 (12.660) | -34.43 (52.810)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 43
  Percent Change at EOT of Cycle 2 | -73.03 (18.304) | -42.38 (42.375)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 33
  Percent Change at EOT of Cycle 3 | -67.01 (24.723) | -44.07 (36.002)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Percent Change at EOT of Cycle 4 | -55.20 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -52.78 (33.033)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Percent Change at EOT of Cycle 5 | -55.42 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -57.42 (34.250)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -52.62 (33.377)
  Percent Change at EOT of Last Cycle | -60.20 (22.297) | -40.89 (55.305)

27. Secondary Outcome: Change From Baseline in Diary PS Caloric Intake at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in diary PS caloric intake at EOT of each cycle during teduglutide treatment was reported. Here, kilo-calories per kilogram per day was abbreviated as (kcal/kg/day).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
kcal/kg/day
  Change at EOT of Cycle 1 | -16.95 (15.141) | -17.40 (13.401)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Change at EOT of Cycle 2 | -10.46 (0.023) | -18.71 (16.722)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Change at EOT of Cycle 3 | -20.77 (0.206) | -22.09 (18.009)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Change at EOT of Cycle 4 | -34.01 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -24.67 (18.859)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Change at EOT of Cycle 5 | -33.68 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -30.20 (13.754)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -34.46 (20.080)
  Change at EOT of Last Cycle | -24.98 (7.540) | -21.13 (18.284)

28. Secondary Outcome: Percent Change From Baseline in Diary PS Caloric Intake at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in diary PS Caloric intake at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
Percent change
  Percent Change at EOT of Cycle 1 | -35.21 (31.088) | -45.91 (35.484)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Percent Change at EOT of Cycle 2 | -14.63 (1.162) | -48.66 (38.282)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Percent Change at EOT of Cycle 3 | -29.03 (2.083) | -46.75 (38.042)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Percent Change at EOT of Cycle 4 | -50.31 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -53.23 (37.611)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Percent Change at EOT of Cycle 5 | -49.81 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -64.30 (30.289)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -50.89 (25.667)
  Percent Change at EOT of Last Cycle | -45.98 (16.836) | -52.02 (41.386)

29. Secondary Outcome: Change From Baseline in Prescribed PS Caloric Intake at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in prescribed PS caloric intake at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 49
kcal/kg/day
  Change at EOT of Cycle 1 | -16.94 (15.187) | -15.80 (17.337)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 42
  Change at EOT of Cycle 2 | -37.91 (38.003) | -16.00 (18.918)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 32
  Change at EOT of Cycle 3 | -44.01 (27.532) | -20.18 (15.633)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4 | -34.59 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -24.48 (15.899)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5 | -34.76 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -27.83 (15.311)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -33.30 (19.205)
  Change at EOT of Last Cycle | -39.68 (21.758) | -18.60 (19.507)

30. Secondary Outcome: Percent Change From Baseline in Prescribed PS Caloric Intake at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in prescribed PS caloric intake at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 49
Percent change
  Percent Change at EOT of Cycle 1 | -34.79 (31.100) | -40.67 (39.607)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 42
  Percent Change at EOT of Cycle 2 | -50.00 (47.944) | -42.75 (45.563)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 32
  Percent Change at EOT of Cycle 3 | -59.00 (32.825) | -44.74 (35.274)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Percent Change at EOT of Cycle 4 | -50.45 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -54.32 (32.153)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Percent Change at EOT of Cycle 5 | -50.69 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -59.49 (30.789)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -50.67 (26.310)
  Percent Change at EOT of Last Cycle | -64.50 (16.117) | -45.84 (42.242)

31. Secondary Outcome: Number of Participants Who Achieved 100% Reduction in Complete Weaning of PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: Number of participants who achieved at least 100% reduction in complete weaning of PS volume at EOT of each cycle during teduglutide treatment was reported.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
Participants
  EOT of Cycle 1 | 0 | 7
  EOT of Cycle 2: number analyzed (Participants) | 2 | 43
  EOT of Cycle 2 | 0 | 8
  EOT of Cycle 3: number analyzed (Participants) | 2 | 33
  EOT of Cycle 3 | 0 | 6
  EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  EOT of Cycle 4 | 0 | 6
  EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  EOT of Cycle 5 | 0 | 6
  EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  EOT of Cycle 6 | 0 | 0
  EOT of Last Cycle | 0 | 10

32. Secondary Outcome: Change From Baseline in Hours Per Day of Diary PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in hours per day of diary PS usage at EOT of each cycle during teduglutide treatment was reported. Hours per day of diary PS was calculated as: Hours per day of actual PS = (sum of hours per day for each day that PS intake data is recorded within the 7 days prior to the visit / number of days that PS hours per day data is recorded as non-zero within the 7 days prior to the visit).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
hours/day
  Change at EOT of Cycle 1 | -0.57 (0.990) | -3.58 (3.750)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Change at EOT of Cycle 2 | -1.71 (2.424) | -3.55 (4.497)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Change at EOT of Cycle 3 | -3.57 (2.222) | -4.19 (5.036)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Change at EOT of Cycle 4 | -4.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -4.83 (5.069)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Change at EOT of Cycle 5 | -4.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -5.64 (5.392)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -5.14 (4.536)
  Change at EOT of Last Cycle | -3.05 (2.700) | -3.89 (4.881)

33. Secondary Outcome: Percent Change From Baseline in Hours Per Day of Diary PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in hours per day of diary PS usage at EOT of each cycle during teduglutide treatment was reported. Hours per day of diary PS was calculated as: Hours per day of actual PS = (sum of hours per day for each day that PS intake data is recorded within the 7 days prior to the visit / number of days that PS hours per day data is recorded as non-zero within the 7 days prior to the visit).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
Percent change
  Percent Change at EOT of Cycle 1 | -4.76 (8.248) | -33.43 (35.645)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Percent Change at EOT of Cycle 2 | -14.29 (20.203) | -34.12 (41.982)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Percent Change at EOT of Cycle 3 | -26.98 (22.448) | -35.11 (41.822)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Percent Change at EOT of Cycle 4 | -22.22 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -40.68 (42.255)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Percent Change at EOT of Cycle 5 | -22.22 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -47.07 (44.248)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -42.86 (37.796)
  Percent Change at EOT of Last Cycle | -21.69 (21.433) | -37.04 (45.049)

34. Secondary Outcome: Change From Baseline in Hours Per Day of Prescribed PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in hours per day of prescribed PS usage at EOT of each cycle during teduglutide treatment was reported. Hours per day of dairy PS was calculated as: Hours per day of actual PS = (sum of hours per day for each day that PS intake data is recorded within the 7 days prior to the visit / number of days that PS hours per day data is recorded as non-zero within the 7 days prior to the visit).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
hours/day
  Change at EOT of Cycle 1 | 0.00 (0.000) | -2.60 (4.279)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 43
  Change at EOT of Cycle 2 | -3.00 (4.243) | -2.78 (5.479)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 33
  Change at EOT of Cycle 3 | -1.00 (1.414) | -2.79 (5.400)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4 | -4.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -3.43 (5.849)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5 | -4.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -3.93 (6.070)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | 0.00 (0.000)
  Change at EOT of Last Cycle | -1.33 (2.309) | -2.58 (5.666)

35. Secondary Outcome: Percent Change From Baseline in Hours Per Day of Prescribed PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in hours per day of prescribed PS usage at EOT of each cycle during teduglutide treatment was reported. Hours per day of dairy PS was calculated as: Hours per day of actual PS = (sum of hours per day for each day that PS intake data is recorded within the 7 days prior to the visit / number of days that PS hours per day data is recorded as non-zero within the 7 days prior to the visit).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 49
Percent change
  Percent Change at EOT of Cycle 1 | 0.00 (0.000) | -21.27 (34.449)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 42
  Percent Change at EOT of Cycle 2 | -16.67 (23.570) | -22.75 (47.101)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 32
  Percent Change at EOT of Cycle 3 | -5.56 (7.857) | -20.64 (40.735)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 26
  Percent Change at EOT of Cycle 4 | -22.22 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -25.47 (43.906)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Percent Change at EOT of Cycle 5 | -22.22 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -32.28 (48.126)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | 0.00 (0.000)
  Percent Change at EOT of Last Cycle | -7.41 (12.830) | -20.91 (47.918)

36. Secondary Outcome: Change From Baseline in Days Per Week of Diary PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in days per week of diary PS usage at EOT of each cycle during teduglutide treatment was reported. Days per week of diary PS was calculated as: Days per week of actual PS = (number of days with non-zero values for PS volume within the 7 days prior to the visit / number of days for which any PS intake data was recorded within the 7 days prior to the visit) * 7.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
Days/week
  Change at EOT of Cycle 1 | -0.33 (0.577) | -1.41 (2.432)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Change at EOT of Cycle 2 | -1.00 (1.414) | -1.76 (2.508)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Change at EOT of Cycle 3 | -1.50 (2.121) | -2.13 (2.756)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Change at EOT of Cycle 4 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -2.36 (2.956)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Change at EOT of Cycle 5 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -2.70 (3.107)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -3.00 (2.646)
  Change at EOT of Last Cycle | -1.00 (1.732) | -2.14 (2.720)

37. Secondary Outcome: Percent Change From Baseline in Days Per Week of Diary PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in days per week of diary PS usage at EOT of each cycle during teduglutide treatment was reported. Days per week of diary PS was calculated as: Days per week of actual PS = (number of days with non-zero values for PS volume within the 7 days prior to the visit / number of days for which any PS intake data was recorded within the 7 days prior to the visit) * 7.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 39
Percent change
  Percent Change at EOT of Cycle 1 | -4.76 (8.248) | -23.40 (39.994)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 38
  Percent Change at EOT of Cycle 2 | -14.29 (20.203) | -29.07 (41.805)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 29
  Percent Change at EOT of Cycle 3 | -21.43 (30.305) | -31.37 (41.530)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 25
  Percent Change at EOT of Cycle 4 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -34.66 (44.475)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 19
  Percent Change at EOT of Cycle 5 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -39.50 (47.024)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -42.86 (37.796)
  Percent Change at EOT of Last Cycle | -14.29 (24.744) | -34.46 (43.755)

38. Secondary Outcome: Change From Baseline in Days Per Week of Prescribed PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in days per week of prescribed PS usage at EOT of each cycle during teduglutide treatment was reported. Days per week of dairy PS was calculated as: Days per week of actual PS = (number of days with non-zero values for PS volume within the 7 days prior to the visit / number of days for which any PS intake data was recorded within the 7 days prior to the visit) * 7
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
Days/week
  Change at EOT of Cycle 1 | -0.33 (0.577) | -1.42 (2.251)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 43
  Change at EOT of Cycle 2 | -1.00 (1.414) | -1.65 (2.399)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 33
  Change at EOT of Cycle 3 | -1.50 (2.121) | -1.85 (2.623)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Change at EOT of Cycle 4 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -2.15 (2.852)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Change at EOT of Cycle 5 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -2.75 (3.041)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Change at EOT of Cycle 6 |  | -3.00 (2.646)
  Change at EOT of Last Cycle | -1.00 (1.732) | -1.92 (2.538)

39. Secondary Outcome: Percent Change From Baseline in Days Per Week of Prescribed PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Percent change from baseline in days per week of prescribed PS usage at EOT of each cycle during teduglutide treatment was reported. Days per week of dairy PS was calculated as: Days per week of actual PS = (number of days with non-zero values for PS volume within the 7 days prior to the visit / number of days for which any PS intake data was recorded within the 7 days prior to the visit) * 7.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 50
Percent change
  Percent Change at EOT of Cycle 1 | -4.76 (8.248) | -23.18 (36.926)
  Percent Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 43
  Percent Change at EOT of Cycle 2 | -14.29 (20.203) | -27.41 (40.209)
  Percent Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 33
  Percent Change at EOT of Cycle 3 | -21.43 (30.305) | -27.58 (40.258)
  Percent Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 27
  Percent Change at EOT of Cycle 4 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -32.12 (43.730)
  Percent Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 20
  Percent Change at EOT of Cycle 5 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -40.86 (46.839)
  Percent Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 3
  Percent Change at EOT of Cycle 6 |  | -42.86 (37.796)
  Percent Change at EOT of Last Cycle | -14.29 (24.744) | -30.71 (40.861)

40. Other Pre Specified Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (GCS) Score at EOT of Each Cycle During Teduglutide Treatment
Description: PedsQL GCS was designed to measure health-related quality of life in pediatric participants and adolescents (2 to 18 years of age). It encompasses 4 dimensions of functioning (physical [8 items], emotional [5 items], social [5 items], school [3 items]). Age groups were: Toddler (2-4 years), Young pediatric (5-7 years), Pediatric (8-12 years), and Teens (13-18 years). Depending on the participant's age, the questionnaire may be completed by parent/caregiver as appropriate. For the Toddler group, the PedsQL GCS consisted of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consisted of 23 items, with a 3-point Likert scale (0, 2, 4) for the young pediatric, and a 5-point Likert scale for the pediatric and teens groups. Scores are transformed on a scale from 0 to 100 where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 42
Score on a scale
  Physical Functioning: Change at EOT of Cycle 1: number analyzed (Participants) | 2 | 41
  Physical Functioning: Change at EOT of Cycle 1 | -21.88 (8.839) | -2.44 (22.323)
  Physical Functioning: Change at EOT of Cycle 2: number analyzed (Participants) | 1 | 34
  Physical Functioning: Change at EOT of Cycle 2 | -18.75 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 4.69 (22.327)
  Physical Functioning: Change at EOT of Cycle 3: number analyzed (Participants) | 1 | 28
  Physical Functioning: Change at EOT of Cycle 3 | -18.75 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -5.80 (27.093)
  Physical Functioning: Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 22
  Physical Functioning: Change at EOT of Cycle 4 | -9.38 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 4.12 (20.872)
  Physical Functioning: Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 11
  Physical Functioning: Change at EOT of Cycle 5 | -15.63 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 4.83 (20.840)
  Physical Functioning: Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0
  Emotional Functioning: Change at EOT of Cycle 1: number analyzed (Participants) | 2 | 41
  Emotional Functioning: Change at EOT of Cycle 1 | -7.50 (10.607) | -2.07 (16.807)
  Emotional Functioning: Change at EOT of Cycle 2: number analyzed (Participants) | 1 | 34
  Emotional Functioning: Change at EOT of Cycle 2 | 5.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 0.88 (15.249)
  Emotional Functioning: Change at EOT of Cycle 3: number analyzed (Participants) | 1 | 28
  Emotional Functioning: Change at EOT of Cycle 3 | -15.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -0.36 (20.680)
  Emotional Functioning: Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 22
  Emotional Functioning: Change at EOT of Cycle 4 | 5.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 1.82 (22.811)
  Emotional Functioning: Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 11
  Emotional Functioning: Change at EOT of Cycle 5 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 1.36 (23.674)
  Emotional Functioning: Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0
  Social Functioning: Change at EOT of Cycle 1: number analyzed (Participants) | 2 | 41
  Social Functioning: Change at EOT of Cycle 1 | -12.50 (17.678) | 0.49 (18.262)
  Social Functioning: Change at EOT of Cycle 2: number analyzed (Participants) | 1 | 34
  Social Functioning: Change at EOT of Cycle 2 | -25.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 5.29 (20.484)
  Social Functioning: Change at EOT of Cycle 3: number analyzed (Participants) | 1 | 28
  Social Functioning: Change at EOT of Cycle 3 | -30.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 2.14 (24.662)
  Social Functioning: Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 22
  Social Functioning: Change at EOT of Cycle 4 | -15.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 3.86 (23.193)
  Social Functioning: Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 11
  Social Functioning: Change at EOT of Cycle 5 | -15.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 2.95 (20.458)
  Social Functioning: Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0
  School Functioning: Change at EOT of Cycle 1: number analyzed (Participants) | 0 | 31
  School Functioning: Change at EOT of Cycle 1 |  | 3.33 (25.111)
  School Functioning: Change at EOT of Cycle 2: number analyzed (Participants) | 0 | 25
  School Functioning: Change at EOT of Cycle 2 |  | 6.93 (27.096)
  School Functioning: Change at EOT of Cycle 3: number analyzed (Participants) | 0 | 20
  School Functioning: Change at EOT of Cycle 3 |  | 1.17 (33.804)
  School Functioning: Change at EOT of Cycle 4: number analyzed (Participants) | 0 | 15
  School Functioning: Change at EOT of Cycle 4 |  | 9.89 (25.233)
  School Functioning: Change at EOT of Cycle 5: number analyzed (Participants) | 0 | 8
  School Functioning: Change at EOT of Cycle 5 |  | 8.33 (23.721)
  School Functioning: Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0

41. Other Pre Specified Outcome: Change From Baseline In PedsQL GCS Score at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 40
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: Analysis was performed using safety population. Here, overall number of participants analyzed refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. Data was collected and analyzed for all the four arms: NTT/NTT, NTT/TED, TED/NTT and TED/TED. Participants who received teduglutide treatment could enter a NT period when the teduglutide treatment criteria were not met.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 4 | 1 | 1 | 14
Score on a scale
  Physical Functioning: Change at Last NT: number analyzed (Participants) | 4 | 1 | 1 | 13
  Physical Functioning: Change at Last NT | 3.91 (10.636) | -3.13 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 31.25 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 13.56 (22.573)
  Emotional Functioning: Change at Last NT | -2.50 (15.546) | -10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 2.50 (23.101)
  Social Functioning: Change at Last NT: number analyzed (Participants) | 4 | 1 | 1 | 13
  Social Functioning: Change at Last NT | 0.00 (4.082) | -10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -10.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 7.31 (16.535)
  School Functioning: Change at Last NT: number analyzed (Participants) | 3 | 0 | 1 | 9
  School Functioning: Change at Last NT | 11.67 (45.369) |  | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 3.89 (25.954)

42. Other Pre Specified Outcome: Change From Baseline In PedsQL Total Family Impact Module Score at EOT of Each Cycle During Teduglutide Treatment
Description: PedsQL Family Impact Module was composed of 36 items comprising Physical Functioning (6 items), Emotional Functioning (5 items), Social Functioning (4 items), Cognitive Functioning (5 items), Communication (3 items), Worry (5 items), Daily Activities (3 items) and Family Relationships (5 items). Total family impact score was calculated as the sum of all the items over the number of items answered on all the scales. Scores are transformed on a scale from 0 to 100 were 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 43
Score on a Scale
  Change at EOT of Cycle 1 | -10.65 (9.326) | 1.55 (15.071)
  Change at EOT of Cycle 2: number analyzed (Participants) | 2 | 34
  Change at EOT of Cycle 2 | -2.78 (3.928) | 4.62 (18.250)
  Change at EOT of Cycle 3: number analyzed (Participants) | 2 | 25
  Change at EOT of Cycle 3 | -5.56 (5.893) | 0.20 (20.861)
  Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 22
  Change at EOT of Cycle 4 | 2.78 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 5.27 (21.637)
  Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 10
  Change at EOT of Cycle 5 | -13.19 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 5.08 (16.152)
  Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0

43. Other Pre Specified Outcome: Change From Baseline In PedsQL Total Family Impact Module Score at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 42
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 3 | 1 | 1 | 15
Score on a scale | -3.47 (10.914) | -27.78 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -12.50 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 6.44 (22.648)

44. Other Pre Specified Outcome: Change From Baseline In PedsQL Gastrointestinal Symptoms Module at EOT of Each Cycle During Teduglutide Treatment
Description: PedsQL Gastrointestinal symptoms module was composed of 58 items, comprised of 10 different symptom scales that assess gastrointestinal symptom-related quality of life: food and drink limits, trouble swallowing, heartburn and reflux, nausea and vomiting, gas and bloating, constipation, blood in poop, and diarrhea. Only the scales of food and drink limits (6 items) and diarrhea (7 items) was used in this study. Sub-scale score was calculated as the sum of the items over the number of items answered in the scale. Scores are transformed on a scale from 0 to 100 were 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, and 6 (Cycles 1, 2, 3, 4, and 5 = 28 weeks, and Cycle 6 = 16 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 2 | 39
Score on a scale
  Food and Drink Limits: Change at EOT of Cycle 1 | -12.50 (17.678) | 1.71 (31.250)
  Food and Drink Limits: Change at EOT of Cycle 2: number analyzed (Participants) | 1 | 31
  Food and Drink Limits: Change at EOT of Cycle 2 | -4.17 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 9.41 (35.583)
  Food and Drink Limits: Change at EOT of Cycle 3: number analyzed (Participants) | 1 | 25
  Food and Drink Limits: Change at EOT of Cycle 3 | -4.17 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 11.83 (36.178)
  Food and Drink Limits: Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 22
  Food and Drink Limits: Change at EOT of Cycle 4 | 12.50 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 18.56 (33.227)
  Food and Drink Limits: Change at EOT of Cycle 5: number analyzed (Participants) | 1 | 10
  Food and Drink Limits: Change at EOT of Cycle 5 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 13.33 (25.215)
  Food and Drink Limits: Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0
  Diarrhea: Change at EOT of Cycle 1: number analyzed (Participants) | 1 | 36
  Diarrhea: Change at EOT of Cycle 1 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 8.56 (21.309)
  Diarrhea: Change at EOT of Cycle 2: number analyzed (Participants) | 1 | 30
  Diarrhea: Change at EOT of Cycle 2 | 0.00 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 10.00 (19.162)
  Diarrhea: Change at EOT of Cycle 3: number analyzed (Participants) | 0 | 23
  Diarrhea: Change at EOT of Cycle 3 |  | 11.49 (23.665)
  Diarrhea: Change at EOT of Cycle 4: number analyzed (Participants) | 1 | 20
  Diarrhea: Change at EOT of Cycle 4 | -3.57 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 8.57 (23.702)
  Diarrhea: Change at EOT of Cycle 5: number analyzed (Participants) | 0 | 9
  Diarrhea: Change at EOT of Cycle 5 |  | 5.56 (27.147)
  Diarrhea: Change at EOT of Cycle 6: number analyzed (Participants) | 0 | 0

45. Other Pre Specified Outcome: Change From Baseline In PedsQL Gastrointestinal Symptoms Module at Last Visit During Non-Teduglutide Treatment (NT)
Description: as for outcome 44
Time Frame: Baseline, Last visit in NT (up to Month 39)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
Number analyzed (Participants) | 4 | 1 | 1 | 12
Score on a scale
  Food and Drink Limits: Change at Last NT | -7.29 (32.698) | -29.17 (NA) — Standard deviation could not be calculated because single participant was analyzed. | -8.33 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 5.35 (34.013)
  Diarrhea: Change at Last NT: number analyzed (Participants) | 4 | 0 | 1 | 10
  Diarrhea: Change at Last NT | -4.46 (4.494) |  | 3.57 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 1.70 (19.555)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to 46 months)
Arm/Group | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) | Non-teduglutide/Teduglutide Treatment (NTT/TED) | Teduglutide /Non-teduglutide Treatment (TED/NTT) | Teduglutide/Teduglutide Treatment (TED/TED)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/1 | 2/50
Serious Adverse Events (participants affected / at risk) | 4/7 | 2/3 | 1/1 | 41/50
Other Adverse Events (participants affected / at risk) | 6/7 | 3/3 | 1/1 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) (N=7) | Non-teduglutide/Teduglutide Treatment (NTT/TED) (N=3) | Teduglutide /Non-teduglutide Treatment (TED/NTT) (N=1) | Teduglutide/Teduglutide Treatment (TED/TED) (N=50)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 16 (31)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 15 (25)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis astroviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malassezia infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Overgrowth bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Astrovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device expulsion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-teduglutide/Non-teduglutide Treatment (NTT/NTT) (N=7) | Non-teduglutide/Teduglutide Treatment (NTT/TED) (N=3) | Teduglutide /Non-teduglutide Treatment (TED/NTT) (N=1) | Teduglutide/Teduglutide Treatment (TED/TED) (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0) | 15 (33)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (10)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 14 (29)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (12) | 3 (11) | 1 (1) | 25 (77)
Catheter site discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site extravasation (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 8 (9)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 16 (21)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Malassezia infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 9 (15)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 5 (9)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (1) | 0 (0) | 15 (41)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (15)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 9 (13)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 5 (11)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (16)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood 25-hydroxycholecalciferol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Gastrointestinal stoma output increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (24)
Lethargy (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 3 (5)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 7 (12)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Learning disability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 16 (41)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 0 (0) | 2 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 10 (26)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 11 (20)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT02954458/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT02954458/SAP_001.pdf